CLINICAL TRIAL: NCT05862909
Title: Efficacy of a Web-Based Emotion Regulation Intervention for Patients With Congenital Heart Disease: A Three-Armed Randomized Clinical Trial
Brief Title: Efficacy of a Web-Based Emotion Regulation Intervention for Patients With Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Competence Network for Congenital Heart Defects (Other Government)
Responsible Party: Principal Investigator, Luise Pruessner, Principal Investigator, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ER-CHD
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Congenital Heart Disease; Emotional Regulation
Keywords: Congenital Heart Disease; Emotional Regulation; Internet-Based Interventions; Emotions
MeSH Terms: conditions — Heart Defects, Congenital; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two intervention groups and a waiting list control group
Who Masked: Investigator, Outcomes Assessor
Masking Description: The group allocation variable will be masked during the data analyses to minimize possible bias concerning the statistical procedure. For this purpose, an independent researcher will delete all information in the dataset indicating the group allocation. Therefore, the evaluator does not know which expression of the group variable represents the CHD-specific intervention, the general intervention, or the waitlist control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (IG 1) (Experimental): CHD-specific web-based emotion regulation intervention
  Interventions: Other: CHD-specific web-based emotion regulation intervention
- Intervention group (IG 2) (Active Comparator): General web-based emotion regulation intervention
  Interventions: Other: General web-based emotion regulation intervention
- Waitlist control group (CG) (No Intervention): 8-week waiting period

INTERVENTIONS:
Other: CHD-specific web-based emotion regulation intervention — CHD-specific web-based emotion regulation intervention with ten video-based sessions covering emotional challenges of CHD and effective emotion regulation strategies (i.e., reappraisal, acceptance, problem solving, distraction, rumination, avoidance, suppression). To integrate the intervention into emotional experiences occurring in the daily life of patients with CHD, the sessions are supported by everyday emotion regulation exercises using an ecological momentary intervention.
  Arms: Intervention group (IG 1)
Other: General web-based emotion regulation intervention — General web-based emotion regulation intervention with ten video-based sessions covering topics related to emotional awareness and effective emotion regulation strategies (i.e., reappraisal, acceptance, problem solving, distraction, rumination, avoidance, suppression). To integrate the intervention into emotional experiences occurring in daily life, the sessions are supported by everyday emotion regulation exercises using an ecological momentary intervention.
  Arms: Intervention group (IG 2)

SUMMARY:
Congenital heart disease (CHD) is associated with daily stressors and functional impairments that can cause negative emotions. Emotion regulation abilities may determine whether people with CHD develop psychopathology or adapt to the illness-related regulatory demands. This three-arm randomized clinical trial evaluates the efficacy of emotion regulation interventions in individuals with CHD.

Patients with CHD over 18 years will be randomly assigned to a CHD-specific web-based emotion regulation intervention, a general web-based emotion regulation intervention, or a waitlist control group with delayed intervention access (8 weeks). The interventions are based on cognitive behavioral therapy, including everyday emotion regulation exercises and psychoeducation via video and audio files. Four and eight weeks after baseline, emotion regulation, well-being, depression, anxiety, perceived stress, life satisfaction, and illness identity will be assessed.

Both interventions are expected to improve emotion regulation abilities, well-being, depressive symptoms, anxiety, perceived stress, life satisfaction, and illness identity four and eight weeks after baseline compared to the waitlist control group. The disease-specific intervention is hypothesized to be superior as it targets everyday emotional problems in CHD patients.

DETAILED DESCRIPTION:
Background: Congenital heart disease (CHD) is associated with significant everyday stressors and impairments in functioning that can induce various negative emotions such as fear, anger, or sadness. When faced with negative emotions caused by the chronic illness, emotion regulation abilities might be central for determining whether individuals with CHD develop symptoms of psychopathology or successfully adjust to the illness-related regulatory demands. Therefore, training emotion regulation abilities offers a promising approach to enhancing psychological well-being in individuals affected by CHD. As patients with CHD face specific challenges, disease-specific emotion regulation interventions may be beneficial in promoting successful adjustment to the condition. Nevertheless, no studies have been conducted to test the effectiveness of emotion regulation interventions for individuals with CHD.

Method: The present three-armed randomized clinical trial evaluates the efficacy of web-based emotion regulation interventions in individuals with CHD. Patients with CHD over 18 years old will be randomly assigned to:

1. A CHD-specific web-based emotion regulation intervention.
2. A general web-based emotion regulation intervention.
3. A waitlist control group with delayed intervention access (8 weeks).

The interventions are conducted via mobile phone or desktop browsers and are based on cognitive behavioral therapy, including everyday emotion regulation exercises and psychoeducation via video material and audio files. Four and eight weeks after baseline, emotion regulation abilities, well-being, depression, anxiety, perceived stress, life satisfaction, and illness identity will be assessed as outcome measures.

Hypotheses: Both interventions are expected to enhance emotion regulation abilities four and eight weeks after baseline compared to the waitlist control group. In addition, the interventions are hypothesized to improve well-being, depressive symptoms, anxiety, perceived stress, life satisfaction, and illness identity. The disease-specific intervention is assumed to be superior to the general emotion regulation intervention as it targets everyday emotional challenges in CHD patients.

ELIGIBILITY:
Inclusion criteria:

* sufficient German language skills (C1)
* permanent internet access during the study period
* diagnosis of a congenital heart disease
* ≥ 18 years of age

Exclusion criteria:

* incapacity to provide informed consent
* acute suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Changes in emotion regulation difficulties | 0 weeks, 4 weeks, 8 weeks
  The Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) consists of 36 items answered on a 5-point scale. The overall score ranges from 36 to 180. Higher values indicate a higher level of emotion regulation difficulties.

SECONDARY OUTCOMES:
Changes in emotion regulation strategy use | 0 weeks, 4 weeks, 8 weeks
  The Heidelberg Form for Emotion Regulation Strategies (HFERST; Izadpanah et al., 2019) consists of 28 items answered on a 5-point scale. For each of the eight emotion regulation strategies (rumination, reappraisal, acceptance, problem solving, suppression of emotional expression, suppression of emotional experience, avoidance, social support), a score ranging from 1 to 5 can be calculated. Higher values indicate a more frequent emotion regulation strategy use.
Changes in well-being | 0 weeks, 4 weeks, 8 weeks
  The World Health Organization Well-Being Index (WHO-5; Topp et al., 2015) consists of 5 items answered on a 6-point scale. The overall score ranges from 0 to 100. Higher values indicate a higher level of well-being.
Changes in depressive symptoms | 0 weeks, 4 weeks, 8 weeks
  The Patient Health Questionnaire (PHQ-9; Kroenke et al., 2001) consists of 9 items answered on a 4-point scale. The overall score ranges from 0 to 27. Higher values indicate a higher level of depressive symptomology.
Changes in anxiety symptoms | 0 weeks, 4 weeks, 8 weeks
  The General Anxiety Disorder Scale (GAD-7; Spitzer et al., 2006) consists of 7 items answered on a 4-point scale. The overall score ranges from 0 to 21. Higher values indicate a higher level of anxiety symptoms.
Changes in perceived stress | 0 weeks, 4 weeks, 8 weeks
  The Perceived Stress Scale (PSS-4; Klein et al., 2014) consists of 4 items answered on a 5-point scale. The overall score ranges from 0 to 16. Higher values indicate a higher level of perceived stress.
Changes in life satisfaction The satisfaction with life scale consists of 5 items answered on a 7-point scale. | 0 weeks, 4 weeks, 8 weeks
  The satisfaction with life scale (SWLS; Diener et al., 1985) consists of 5 items answered on a 7-point scale. The overall score ranges from 5 to 35. Higher values indicate a higher life satisfaction.
Changes in illness identity | 0 weeks, 4 weeks, 8 weeks
  The Illness Identity Questionnaire (IIQ; Oris et al., 2016) consists of 25 items answered on a 5-point scale. The overall score ranges from 25 to 125. Higher values indicate a higher level of perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Luise Pruessner, Principal Investigator — Department of Psychology, Heidelberg University, Heidelberg (Germany); Steffen Hartmann, Principal Investigator — Department of Psychology, Heidelberg University, Heidelberg (Germany); Anna-Lena Ehmann, Principal Investigator — Department of Psychology, Heidelberg University, Heidelberg (Germany); Sven Barnow, Principal Investigator — Department of Psychology, Heidelberg University, Heidelberg (Germany); Ulrike Bauer, Principal Investigator — National Register for Congenital Heart Defects, Berlin (Germany); Paul Helm, Principal Investigator — National Register for Congenital Heart Defects, Berlin (Germany)
Locations (1):
- Competence Network for Congenital Heart Defects, Berlin, Germany

REFERENCES:
- [Background] Izadpanah S, Barnow S, Neubauer AB, Holl J. Development and Validation of the Heidelberg Form for Emotion Regulation Strategies (HFERST): Factor Structure, Reliability, and Validity. Assessment. 2019 Jul;26(5):880-906. doi: 10.1177/1073191117720283. Epub 2017 Jul 21. PMID 28730850
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Oris L, Rassart J, Prikken S, Verschueren M, Goubert L, Moons P, Berg CA, Weets I, Luyckx K. Illness Identity in Adolescents and Emerging Adults With Type 1 Diabetes: Introducing the Illness Identity Questionnaire. Diabetes Care. 2016 May;39(5):757-63. doi: 10.2337/dc15-2559. Epub 2016 Mar 17. PMID 26989179
- [Background] Klein EM, Brahler E, Dreier M, Reinecke L, Muller KW, Schmutzer G, Wolfling K, Beutel ME. The German version of the Perceived Stress Scale - psychometric characteristics in a representative German community sample. BMC Psychiatry. 2016 May 23;16:159. doi: 10.1186/s12888-016-0875-9. PMID 27216151
- [Background] Ritschel LA, Tone EB, Schoemann AM, Lim NE. Psychometric properties of the Difficulties in Emotion Regulation Scale across demographic groups. Psychol Assess. 2015 Sep;27(3):944-54. doi: 10.1037/pas0000099. Epub 2015 Mar 16. PMID 25774638
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Derived] Pruessner L, Hartmann S, Ehmann AL, Barnow S, Bauer UMM, Helm PC. Digital Emotion Regulation Interventions for Patients With Congenital Heart Disease: A Randomized Clinical Trial. JAMA Netw Open. 2025 Oct 1;8(10):e2538813. doi: 10.1001/jamanetworkopen.2025.38813. PMID 41134574